CLINICAL TRIAL: NCT03284658
Title: BioTyrosin - Biomarker for the Early Diagnosis and Monitoring in Tyrosinemia Type 1 - An International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for the Early Diagnosis and Monitoring in Tyrosinemia Type 1 (BioTyrosin)
Acronym: BioTyrosin
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BTY 06-2018
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Tyrosinosis; Hepatorenal Tyrosinemia; Fumarylacetoacetase Deficiency; Fah Deficiency; Metabolic Disorders
Keywords: Tyrosinemia Type 1; Biomarker
MeSH Terms: conditions — Tyrosinosis; Tyrosinemias; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectrometry, a blood sample of maximal 7,5 ml blood will be taken from the patient via using a dry blood spot filter card. To proof the correct diagnosis a Tyrosinemia type 1, in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of a Tyrosinemia type 1 will be done.
  The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with a Tyrosinemia type 1 or high-grade suspi-cion for Tyrosinemia type 1

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Tyrosinemia type 1 from blood (plasma)

DETAILED DESCRIPTION:
Hereditary Tyrosinemia type 1 (HT-1) is a rare genetic disorder in which the newborn child lacks the ability to break down the amino acid tyrosine. As a result of this deficiency, toxic sub-stances build up in the blood and can cause liver failure, kidney dysfunction and neurological problems. There are two different forms of the disease - acute and chronic. The acute form is most common.

Worldwide, Tyrosinemia type 1 affects about one newborn child in 100,000, although geo-graphical variation is seen.

Tyrosinemia type 1 is hereditary. The disorder is caused by a defect in the gene coding for the enzyme responsible for breaking down tyrosine. For a child to be affected by the disease, both parents have to carry a defective gene. The risk of being born with Tyrosinemia type 1, i.e. receiving both genes from the parents, is thus 25%.

Children with Tyrosinemia type 1 can display symptoms such as failure to gain weight and grow at the expected rate, diarrhea, vomiting, enlarged liver, liver failure, accumulation of fluid in the peritoneal cavity, kidney failure, softening of the bones (rickets) and liver tumors.

The acute form usually appears in the first few months of life. The child has a slow weight gain plus fever, diarrhea, blood in the feces and vomiting. The liver is enlarged and yellowing of the skin and the whites of the eyes (jaundice) with an increased tendency to bleed (particularly nosebleeds) may be evident. The spleen and abdomen can also be enlarged and the legs swollen. Without treatment, liver failure and clotting problems can arise.

Children with the chronic form of Tyrosinemia type 1 develop symptoms gradually. The child can suffer from enlarged liver, distended abdomen (due to enlarged liver and spleen, acites and excessive fluids), changes in skeleton, and liver and kidney failure. Symptoms such as abdominal pain, damage to the peripheral nerves and high blood pressure appear. In addition, symptoms common in acute intermittent porphyria can also occur. If the child is not treated, it will develop liver failure and liver tumors.

The condition is also referred to as hepatorenal Tyrosinemia, and is the most critical variant of Tyrosinemia. The main function of the FAH gene is to regulate the production of the enzyme fumarylacetoacetase that is required to break down or metabolize amino acid tyrosine. The mutations of FAH gene leads to a deficiency of the enzyme fumarylacetoacetase, which then leads to a failure in breaking down tyrosine.

Tyrosinemia type 1 is suspected on the basis of clinical presentation. Diagnostic investigations include analyses of amino acids, succinylacetone and alpha-fetoprotein.

Today, the condition can be treated by diet, medication and liver transplantation. Liver trans-plantation was once the only treatment, but since a new drug was introduced in 1991, survival has increased significantly. Nevertheless, diet and special protein replacements remain an important part of life-long treatment.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the dis-ease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of Tyrosinemia type 1 or a high-grade suspicion for Tyrosinemia type 1

High-grade suspicion present, if one or more inclusion criteria are valid:

* Positive family anamnesis for Tyrosinemia type 1
* Hepatomegaly
* Splenomegaly
* Ascites
* Coagulopathy

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Tyrosinemia type 1 or no valid criteria for profound suspicion of Tyrosinemia type 1

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a Tyrosinemia type 1 or high-grade suspi-cion for Tyrosinemia type 1
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Tyrosinemia Type 1 disease related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the FAH gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Tyrosinemia type 1 specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (3):
- Centogene AG, Rostock, Germany
- NIRMAN Navi Mumbai Institute of Research In Mental And Neurological Handicap/Pediatric Geneticist, Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided